CLINICAL TRIAL: NCT06368804
Title: Comparison of Two Antibiotic Regimens for the Treatment of Early Airways Infection With Pseudomonas Aeruginosa in Adults With Bronchiectasis: a Non-inferiority Randomized Controlled Trial.
Brief Title: Comparison of Two Antibiotic Regimens for the Treatment of Early Airways Infection With PA in Adults With Bronchiectasis
Acronym: ANTEIPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANTEIPA; 2022-A01575-38 (Other: ID-RCB)
Record Dates: First submitted 2024-02-22; First posted 2024-04-16 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Bronchiectasis
Keywords: Non cystic fibrosis bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral fluoroquinolone + nebulized colistimethate sodium (Experimental)
  Interventions: Drug: Antibiotic monotherapy treatment and follow-up
- IV beta-lactam antibiotic (ceftazidime) + oral fluoroquinolone + nebulized colistimethate sodium (Active Comparator)
  Interventions: Drug: Antibiotic bitherapy treatment and follow-up

INTERVENTIONS:
Drug: Antibiotic monotherapy treatment and follow-up — 1. a 3-months treatment period, including:
     * an initial phase of 14 days, combining an oral fluoroquinolone (ciprofloxacin 750mg tw/d) with nebulized sodium colistimethate (1 Million Units tw/d)
     * a maintenance phase of 2.5 months: nebulized sodium colistimethate (1 MU tw/d) ;
  2. a subsequent follow-up period of 9 months (i.e. until 12 months after the start of antibiotic therapy against Pseudomonas aeruginosa).
  Arms: Oral fluoroquinolone + nebulized colistimethate sodium
Drug: Antibiotic bitherapy treatment and follow-up — 1. a 3-months treatment period, including:
     * an initial phase of 14 days, combining an IV beta-lactam antibitic (ceftazidime 4 or 6g/d) and an oral fluoroquinolone (ciprofloxacin 750mg tw/d) with nebulized sodium colistimethate (1 Million Units tw/d)
     * a maintenance phase of 2.5 months: nebulized sodium colistimethate (1 MU tw/d) ;
  2. a subsequent follow-up period of 9 months (i.e. until 12 months after the start of antibiotic therapy against Pseudomonas aeruginosa).
  Arms: IV beta-lactam antibiotic (ceftazidime) + oral fluoroquinolone + nebulized colistimethate sodium

SUMMARY:
Chronic airways infection with Pseudomonas aeruginosa (PA) is associated with increased frequency of exacerbations, deterioration in quality of life and increased mortality in adult patients with bronchiectasis. Current guidelines suggest the prescription of an eradication antibiotic treatment for a first episode of PA infection (early PA infection). Several antibiotic regimens may be proposed, ranging from a monotherapy with oral fluoroquinolone (FQ) to an intravenous cotherapy with the addition of inhaled antibiotics that seems to improve the rate of PA eradication. As no study strictly favoured one regimen, current practices are heterogeneous and could certainly benefit from stronger evidence, with both medical and economic impact.

DETAILED DESCRIPTION:
According to current knowledge, the early combination of an oral FQ to an inhaled antibiotic could be an acceptable alternative to a systemic cotherapy. Indeed, such regimen allows avoiding IV drugs use, facilitating ambulatory management and influencing patient's quality of life and costs, and may achieve similar PA-eradication rate.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosis of bronchiectasis on thoracic CT-scan
* Recent isolation of P. aeruginosa (PA) in a respiratory sample (spontaneous or induced sputum or other lower respiratory tract sample obtained by bronchoscopy) within the last 3 months, with a PA positive respiratory sample obtained ≤ 3 weeks before randomization
* Patient either Pseudomonas naive (i.e., never previously isolated PA) or Pseudomonas free (i.e., infection-free for ≥1 year, proven by at least two PA negative respiratory sample during the last year)
* Patient affiliated with the French health care system
* Able to understand and sign a written informed consent form

Exclusion Criteria:

* Confirmed diagnosis of cystic fibrosis
* Pregnancy or breastfeeding
* Women of childbearing potential (after the first menstrual period and until menopause or permanent sterility (hysterectomy, bilateral salpingectomy and bilateral oophorectomy)) who refuse to use effective contraception (hormonal or mechanical) for 3 months and/or to undergo pregnancy tests at baseline, 1 month and 3 months after baseline.
* Isolation of PA in a respiratory specimen (spontaneous or induced sputum or other lower respiratory tract specimen obtained by bronchoscopy) more than 3 months to 12 months prior to randomization.
* PA resistant to ciprofloxacin or ceftazidime
* Severe exacerbation requiring admission to an intensive care unit (e.g. for non-invasive ventilatory support, invasive mechanical ventilation, catecholamine or any other organ supportive therapy)
* Prior severe reaction, hypersensitivity reaction or other contraindication to any of the treatments in study (ciprofloxacin, beta-lactam, colistimethate sodium)
* Prior severe bronchospasm attributed to a nebulization
* Patients already receiving PA suppressive therapy with an inhaled antibiotic (long-term azithromycin therapy accepted)
* Prior PA-eradication antibiotic treatment (systemic antibiotic(s) active against PA for ≥ 14 days or nebulized anti-PA antibiotic) within the last year
* Antibiotic treatment active against PA (anti-PA beta-lactam antibiotic and/or FQ and/or aminoglycoside) for more than 3 days before randomisation
* Active cancer or haematological malignancy under active therapy
* Systemic corticosteroid therapy ≥ 20 mg/d. prednisone equivalent for a predictable duration > 4 weeks
* Non-tuberculous mycobacterial infection or positive non-tuberculous mycobacterial respiratory specimen within 1 year prior to inclusion
* Severe chronic renal failure defined by a creatinine clearance (Cockcroft or MDRD) ≤ 30 mL/min/1.73m2 or chronic haemodialysis
* Severe hepatic impairment
* Long-term oxygen therapy and/or noninvasive mechanical ventilation for chronic respiratory insufficiency (except continuous positive airway pressure for OSA) and/or forced expiratory volume at one second (FEV1) <25% of predicted value.
* Patient participating to another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
PA-eradication rate | 6 months
  PA-eradication rate 6 months after the start of antibiotic therapy targeting PA, where PA eradication is defined as follows:
  * Sputum culture (or lower airway specimen culture, if respiratory exacerbation* with inability to perform good quality sputum analysis) negative for PA at the 6-month follow-up visit, or
  * Inability to spit in the absence of a pulmonary exacerbation*, AND
  * No sputum culture or lower airway specimen positive for PA between D90 of antibiotic treatment and the 6-month follow-up visit, in the absence of new antibiotic therapy targeting PA.

SECONDARY OUTCOMES:
Time to first exacerbation | 3, 6 and 12 months-follow up visit, or additional visit
  exacerbation assessment at each follow-up visit, with time (in days) between the start of antibiotic therapy against PA and first exacerbation
1 year-exacerbation rate | 3, 6 and 12 months-follow up visit
  exacerbation assessment at each follow-up visit
Quality-of-life using questionnaires | Inclusion, 3 and 12 months-follow up visit
  Quality of Life-Bronchiectasis (QOL-B)
Quality-of-life using questionnaires | Inclusion, 3 and 12 months-follow up visit
  Bronchiectasis Impact Measure (BIM)
Treatment burden assessment using questionnaires | Inclusion, 3 and 12 months-follow up visit
  Treatment Burden Questionnaire (TBQ)
Quality-of-life using questionnaires | Inclusion, 3 and 12 months-follow up visit
  EQ-5D-5L questionnaire for the medico-economic analysis
Detection of PA at 3-month and 1 year | 3 and 12 months-follow up visit
  Sputum (or lower respiratory tract sample, if clinically justified) culture growing PA
Time to first PA-recurrence | 3, 6 and 12 months-follow up visit
  PA-recurrence in sputum (or lower respiratory tract sample, if clinically justified), with time (in days) between the start of antibiotic therapy against PA and first PA-recurrence
Emergence of FQ-resistant strains of (PA or other bacteria) | 3, 6 and 12 months-follow up visit
  analysis of PA (or other bacteria) susceptibility to ciprofloxacin, if growing on respiratory sample(s) performed between 3 months and 12 months
Adverse event (AE) and serious AE at 12 months follow-up | during the 12 months follow-up
  AE and serious AEs will be recorded during medical interviews and by self-report in the study booklet during the study
Number of premature ending of one of the treatment in study due to any AE | 1 months and 3 months-follow up visit
  Compliance to treatment and AEs will be recorded during medical interviews and by self-report in the study booklet during the study treatment period, time (in days)
Number of premature ending of one of the treatment in study | 1 months and 3 months-follow up visit
  Compliance to treatment will be recorded during medical interviews and by self-report in the study booklet during the study treatment period, time (in days)
Proportion of non-administered doses of nebulized colistin | 1 months and 3 months-follow up visit
  Compliance to treatment will be recorded during medical interviews and by self-report in the study booklet during the study treatment period, time (in days)
Cost and incremental cost effectiveness ratio at 1 year | Inclusion and each follow up visit up to one year for quality of life measures; initial discharge and subsequent exacerbation-related readmissions up to one year.
  Total cost in each group
Cost and incremental cost effectiveness ratio at 1 year | Inclusion and each follow up visit up to one year for quality of life measures; initial discharge and subsequent exacerbation-related readmissions up to one year.
  Total quality adjusted life years (QALYs) in each group
Cost and incremental cost effectiveness ratio at 1 year | Inclusion and each follow up visit up to one year for quality of life measures; initial discharge and subsequent exacerbation-related readmissions up to one year.
  Difference in costs /difference in QALYs

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Amiens-Picardie, Amiens
  - CHU Haut Leveque, Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - CH Pontoise, Cergy-Pontoise
  - Centre hospitalier intercommunal de Créteil, Créteil
  - APHP, Henri Mondor, Créteil
  - Hôpital de la Croix Rousse, HCL, Lyon, Lyon
  - Clinique St Joseph, Marseille
  - CHU Nantes, Nantes
  - CHU H. Pasteur, Nice, Nice
  - Hôpital Pitié Salpêtrière, Paris
  - APHP, Cochin, Paris
  - APHP, Saint Louis, Paris
  - APHP, Tenon, Paris
  - Hôpital Foch, Suresnes, Suresnes
  - CHU H. Larrey, Toulouse, Toulouse
  - CH Versailles, Versailles
  - CH Villefranche s/Saône, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No